CLINICAL TRIAL: NCT05456945
Title: Comparison of the Efficacy of Shotblocker and Acupressure in Reducing Pain Due to Intramuscular Injection in the Emergency Department: A Single-Blind, Randomized Controlled Study
Brief Title: Comparison of the Efficacy of Shotblocker and Acupressure in Reducing Pain Due to Intramuscular Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tülay KILINÇ, Principal İnvestigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: tulay23
Record Dates: First submitted 2022-07-10; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Acute Pain; İnjection; Acupressure; Alternative Medicine
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure (Experimental): Before the injection, patients will be asked to lie in the prone position. The acupressure point (UB32) will be located on the side to be injected. The UB32 point is located in the sacrum region, below the medial and posterior superior iliac spine, in the second sacral foramen. The acupressure point UB32 will be pressed circularly with a stopwatch for 1 minute. Then the acupressure point will be pressed three times in sequence with the thumb directly (pressure equal to 4.5 kg/cm2). Diclofenac sodium (75mg/3ml) will be injected after acupressure.
  Interventions: Other: acupressure application
- Shotblocher (Experimental): Before the injection, patients will be asked to lie in the prone position. The protruding surface of the Shotblocker will be placed in the area just before the injection so that the point of entry with the needle will not be contaminated. Pressure will be applied by keeping the Shotblocker constant throughout the process. The injector will be quickly inserted through the gap in the middle of the shortblocher. Shotblocker will be removed after drug administration.
  Interventions: Device: Shotblocher
- Control group (No Intervention): No intervention will be applied before the injection

INTERVENTIONS:
Other: acupressure application — Acupressure will be applied to the UB32 point
  Arms: Acupressure
Device: Shotblocher — Shotblocher will be administered during injection
  Arms: Shotblocher

SUMMARY:
Various non-pharmacological approaches are used in the relief of pain caused by intramuscular injection. Shotblocher and acupressure, which are among these methods, are easy to apply.More evidence-based studies are needed to fully understand the effectiveness of acupressure an d shotblocher in reducing pain associated with intramuscular injection.This study will be conducted to compare the effectiveness of shotblocker and acupressure in reducing pain associated with intramuscular injection in the emergency department.

DETAILED DESCRIPTION:
Intramuscular injection is a nursing practice that is frequently used in clinical practice. If intramuscular injection is not performed with correct and appropriate methods, it can cause serious complications. These complications include pain, cellulitis, muscle fibrosis and contracture, sterile abscesses, tissue necrosis, granuloma, intravascular injection, hematoma, and nerve injuries. Although it has healing and therapeutic properties, intramuscular injection can cause pain and discomfort in the patient. Intramuscular injection pain develops due to the mechanical trauma caused by the needle entry and the sudden pressure created when the drug is injected into the muscle. Nurses play an active role in eliminating or reducing the pain that occurs in this process. Pharmacological and non-pharmacological methods are used to reduce pain associated with intramuscular injection. Topical anesthetics, one of the pharmacological methods, are limited in use in emergency services due to their slow analgesic effects, risk of systemic toxicity and local side effects. There are various non-pharmacological methods applied to control pain caused by injection. One of the non-pharmacological methods applied to reduce the pain experienced during intramuscular injection is Shotblocker application. It is reported that ShotBlocker reduces pain by temporarily blocking the peripheral nerve endings by preventing the perception of pain and its transmission to the central nervous system. Another method used to reduce pain due to injection is acupressure. Experimental and clinical evidence suggests that acupressure may relieve pain and promote relaxation. In addition, this non-invasive application involves minimal risk and can be easily integrated into the application. Acupressure points such as UB31, UB32, UB33 and UB34 are stated to be beneficial for low back pain, hernia, dysmenorrhea, dysuria, pain. Of these, UB32 and UB31 are clinically frequently used acupressure points. In this study, the UB32 acupressure point will be used to reduce the pain associated with multiple injections.

ELIGIBILITY:
Inclusion Criteria:

* Those who are admitted to the emergency room for the administration of prescription drugs or those who are planned to be injected intramuscularly by the emergency room physician
* Diclofenac sodium (75 mg/3 ml) was ordered to the patient in the emergency department.
* 18 years and older
* Patients who have not had an injection in the same area in the last 2 week
* Having no problems with vision and hearing
* Does not have a disease that can cause loss of sensation and sensory loss
* Open to communication and cooperation
* Patients willing to participate in the study will be included in the study.

Exclusion Criteria:

* Those who apply to the emergency department with complaints of anxiety or trauma (soft tissue traumas, multiple traumas due to traffic accidents or falls, or bone fractures),
* Those who experience a change in consciousness,
* Patients with clinical conditions that require urgent intervention,
* Infection at the injection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 2 minutes
  The visual analog scale will be used to assess the patient's pain intensity. It is a self-reported scale in the form of a 10-cm ruler indicating no pain at one end and unbearable pain at the other. Accordingly, the patient is told to evaluate his/her pain between 0 and 10, with 0 indicating "no pain" and 10 indicating "unbearable pain
Verbal category scale | 2 minutes
  The verbal category scale is a one-dimensional, simple, descriptive scale. Patients are asked to state the most appropriate word to describe their pain while filling in the scale. To describe the severity of pain, the patients had to choose from among (1) mild, (2) disturbing, (3) severe, (4) very severe, and (5) unbearable 5. The verbal category scale is a one-dimensional, simple, descriptive scale. Patients are asked to state the most appropriate word to describe their pain while filling in the scale. To describe the severity of pain, the patients had to choose from among (1) mild, (2) disturbing, (3) severe, (4) very severe, and (5) unbearable